CLINICAL TRIAL: NCT05923905
Title: Randomized Double-blind Controlled Exploratory Clinical Study to Evaluate the Efficacy and Safety of FB1006 in the Treatment of ALS Patients
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of FB1006 in the Treatment of ALS Patients
Acronym: FB1006
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M2022300
Record Dates: First submitted 2023-02-06; First posted 2023-06-28 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-01

CONDITIONS: Sporadic and Familial Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FB1006 test group (Experimental): Take FB1006 at night,30mg/day
  Interventions: Drug: FB1006
- placebo group (Placebo Comparator): Take placebo at night,30mg/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FB1006 — 30mg/day
  Arms: FB1006 test group
Drug: Placebo — 30mg/day
  Arms: placebo group

SUMMARY:
This is a randomized double-blind controlled exploratory clinical study to evaluate the efficacy and safety of FB1006 in the treatment of amyotrophic lateral sclerosis (ALS) patients.

DETAILED DESCRIPTION:
This is a randomized double-blind controlled exploratory clinical study to evaluate the efficacy and safety of FB1006 in the treatment of amyotrophic lateral sclerosis (ALS) patients. The study has two phases: the first phase is 24 weeks, using a randomized double-blind placebo-controlled design; the second phase is 24 weeks, using an open-label study design. FB1006 was approved by the National Medical Products Administration（NMPA）on June 21, 2021.

ELIGIBILITY:
Inclusion Criteria:

1. World Federation of Neurology modified El Ecorial criteria for diagnosis of patients with laboratory support probable, clinically probable, or definite sporadic and familial amyotrophic lateral sclerosis (ALS)
2. Age 18 to 80 years old
3. ALS duration no longer than 18 months(from day of onset)
4. Patient 's ALSFRS-R total scored ≥27，Each single item is scored at least 2（dyspnoea, orthopnea and respiratory insufficiency ≥3）
5. Forced vital capacity (FVC%) no less than 70% of predicted normal for gender, height and age
6. According to brain function AI analysis in accordance with depressive EEG characteristics
7. Women and men of childbearing potential should use medically acceptable contraception
8. Voluntarily participate, and sign an informed consent form

Exclusion Criteria:

1. Patients with dementia or severe neurological, psychiatric or systemic disease that is poorly controlled or may interfere with the conduct of the trial or the results of the trial
2. Pregnant women and lactating women
3. Suicide attempt or attempted suicide
4. Combined with other neurological diseases similar to ALS symptoms, or affecting the evaluation of drug efficacy, such as cervical spondylotic myelopathy, lumbar spondylosis, dementia, etc.
5. Patients with history of spinal surgery after ALS onset
6. ALT or AST > 2 times ULN，creatinine clearance < 60 mL/min/1.73m2 (MDRD)
7. Patients who are allergic to the investigational product
8. Having participated in other clinical studies within 3 months before randomization
9. Patients that the investigator considers unsuitable for participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
ROADS (Rasch-Built Overall Amyotrophic Lateral Sclerosis Disability Scale) Score | 24 weeks
  Changes in ROADS from baseline to 24 weeks. ROADS score ranges from 0 to 56 points, and higher scores indicate better basic daily function.

SECONDARY OUTCOMES:
ALSFRS-R (Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised) Score | 24 weeks
  Changes in ALSFRS-R from baseline to 24 weeks. ALSFRS-R score ranges from 0 to 48 points, and higher scores indicate milder functional impairment.
ALSFRS-R Score | 12 weeks, 36 weeks, and 48 weeks
  Changes in ALSFRS-R and slope of score decrease during the observation period. ALSFRS-R score ranges from 0 to 48 points, and higher scores indicate better function.
ROADS (Rasch-Built Overall Amyotrophic Lateral Sclerosis Disability Scale) Score | 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 28 weeks, 32 weeks, 36 weeks, 40 weeks, 44 weeks, and 48 weeks
  Changes in ROADS during the observation period. ROADS score ranges from 0 to 56 points, and higher scores indicate better basic daily function.
ALSAQ-40 (Amyotrophic Lateral Sclerosis Assessment Questionnaire-40) Score | 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Changes in ALSAQ-40 during the observation period. ALSAQ-40 score ranges from 0 to 160 points, and higher scores indicate better quality of life.
Zung 's Self-Rating Depression Scale | 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 28 weeks, 32 weeks, 36 weeks, 40 weeks, 44 weeks, and 48 weeks.
  Changes in Zung 's score during the observation period. Zung 's score ranges from 0 to 100 points, and higher scores indicate more severity of depression.
Metabolic Level | 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
  Changes in metabolic equivalent (MET) value during the observation period. MET is measured by cardiopulmonary exercise test (CPET).
FVC% (Forced Vital Capacity) | 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
  Changes in FVC% during the observation period.
Body Weight | 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
  Changes in body weight during the observation period.
MRC (Medical Research Council) Scale | 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
  Changes in MRC classification during the observation period. MRC ranges from 0 to V grades, and higher grades indicate higher muscle strength.
MUNIX (Motor Unit Number Index) | 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
  Changes in MUNIX during the observation period. MUNIX is obtained from electromyography (EMG) in terms of quadriceps, deltoid, abductor digiti minimi (ADM), and tibialis anterior (TA) muscles.
Language Disorders | 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
  Occurrence of language disorders during the observation period. Language disorders is detected by AI (Artificial Intelligence) analysis from wearable electroencephalographic device.
Hand Delicate Function | 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
  Changes in hand delicate function during the observation period. Hand delicate function is detected by AI (Artificial Intelligence) analysis from wearable electromyographic device.

OTHER OUTCOMES:
Important Events in ALS Progression | 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
  Occurrence of important events in ALS Progression, include indwelling gastric tube/gastrostomy, respiratory support, death, etc.
ESS (Epworth Sleepiness Scale) Score | 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
  Changes in ESS score during the observation period. ESS score ranges from 0 to 24 points, and higher scores indicate more severity of daytime somnolence.
PSQI (Pittsburgh Sleep Quality Index) Score | 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
  Changes in PSQI during the observation period. PSQI score ranges from 0 to 21 points, and higher scores indicate poorer sleep quality.
Biomarkers | 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
  Changes in serum NFL, BDNF, GDNF, inflammatory factors (TNF, IL-1, IL-6, IL-18, CRP) during the observation period.
EEG (Electroencephalogram) | 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
  Occurrence of clinically significant abnormalities during the observation period.
CMAP (Compound Muscle Action Potential) | 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
  Changes in CMAP during the observation period. CMAP is obtained from electromyography (EMG) in terms of medianus, peroneus, radialis, tibialis, and ulnaris muscles.
Adverse Events | 48 weeks
  Occurrence of any adverse events and clinically significant laboratory abnormalities during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Fan DongSheng, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No